CLINICAL TRIAL: NCT03527407
Title: MIDAS: Minimal-dataset for the Assessment of Surgical Outcomes - Potential in Hip Surgery (ch18Jakob3)
Brief Title: MIDAS: Minimal-dataset for the Assessment of Surgical Outcomes - Potential in Hip Surgery
Acronym: MIDAS
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-00763; ch18Jakob3
Record Dates: First submitted 2018-04-16; First posted 2018-05-17 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Hip Injuries
MeSH Terms: conditions — Hip Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Swiss legislation requires health service providers to collect such information. of medical quality indicators as part of the quality and performance audit (Article 22a KVG). In addition, comparisons of clinics or specialist specialists on cost and quality of results are required (Art. 49 (8)).

Currently, the quality of a medical therapy is evaluated rather negatively on the absence (or occurrence) of complications. In contrast, however, the goal of therapy must be to improve or maintain the health-related quality of life (HRQoL). Accordingly, the Swiss Society of Surgery (SGC-SSC), in collaboration with the Association for Quality Assurance in Surgery (AQC), has developed a minimum dataset designed to assess the quality of life of patients after surgical intervention. In order to enable Switzerland to be comparatively independent of the discipline, generic (in the Research Plan - MIDAS -V2, date 24.05.2017 Page 5/57 Contrary to disease-specific) survey instruments proposed that cover the general quality of life in its different facets, regardless of the function of individual organ systems. The complication documentation was not completely abandoned in this proposal, but is only a quality indicator among many due to patient-related outcome measurements.

However, the development of a minimal data set with quality indicators that are applicable across all surgical sub-disciplines for evaluating the quality of treatment of acute and chronic diseases raises a number of fundamental questions that can only be answered to a limited extent without empirical studies. Five essential questions are:

I. Is it sufficient to work with generic quality of life tools or is it necessary to use disease / indication specific instruments or functional tests? II. Which is the best, solid time for a follow-up? III. Is it possible and useful to make a third-party determination of the quality of life in patients with limited cognitive abilities? IV. Which preoperative risk factors should be documented so that sufficient adjustment for case mix differences in hospital comparisons can be made? V. Which perioperative and postoperative factors, in particular complications, must be raised beyond the quality of life, as they reflect an independent aspect of quality?

ELIGIBILITY:
Inclusion Criteria:

- Standard therapy of one of the following diagnoses

* Femoral neck fracture after low-energy trauma (implantation of a head endoprosthesis)
* Coxarthrosis (implantation of a total hip prosthesis)

Exclusion Criteria:

* Rejection of study participation or standard therapy
* Patients who are unlikely to attend routine follow-up (e.g., tourists)
* Patients in palliative care
* Malignancy (known or diagnosed in the course of time)
* Patients with a limited knowledge of German, who can answer the questionnaire even with the help of a study nurse seems unrealistic
* Participation in an interfering clinical intervention study within the last three months
* persons unable to consent (long-term incapacity to consent)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The current study has been designed to support decisions on how to define a minimal data set and how to organize data collection to obtain valid data. Two patient groups will serve as an example:
  1. patients with arthritis of the hip joint and indication for total prosthetic joint replacement surgery
  2. patients with acute femoral neck fracture and indication for partial or total prosthetic joint replacement surgery
Sampling Method: Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-01-06 (Actual); Study Completion 2021-01-06 (Actual)

PRIMARY OUTCOMES:
Changes to Baseline in the generic scores EuroQuol5 (EQ-5D) | baseline, month 3 and month 12
  The degree of mapping the influence of known factors for the quality of therapy to changes to Baseline in the generic scores EuroQuol5 (EQ-5D).
  different measuring times between 3 and 12 months.
Changes to Baseline in the Health Utility Index Mark 3 (HUI3) | baseline, month 3 and month 12
  The degree of mapping the influence of known factors for the quality of therapy to changes to Baseline in the Health Utility Index Mark 3 (HUI3).
  different measuring times between 3 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Jakob, Prof MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Department of Orthopedic and Trauma Surgery, University Hospital Basel, Basel, Switzerland